CLINICAL TRIAL: NCT02326415
Title: Prospective Randomised Study Comparing Clinical Pathway With "Fast-Track" Versus Usual Protocol In Uncomplicated Acute Appendicitis
Brief Title: Clinical Pathway With "Fast-Track" In Uncomplicated Acute Appendicitis
Acronym: CLIPUA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Jesus Abrisqueta Carrion, Ph D, Hospital Universitario Virgen de la Arrixaca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCUVA-CPA-JAC
Record Dates: First submitted 2014-12-15; First posted 2014-12-29 (Estimated); Last update posted 2014-12-29 (Estimated); Status verified 2014-12

CONDITIONS: Uncomplicated Acute Appendicitis
Keywords: Acute Appendicitis; Appendectomy; Fast-Track; Clinical Pathway
MeSH Terms: conditions — Appendicitis | interventions — Critical Pathways

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinical Pathway With "Fast-Track" (Active Comparator): All the clinical performances that the health personal have to do about the patient with uncomplicated acute appendicitis is already established in a care maps since the patient comes to hospital until the discharge.
  Interventions: Other: Clinical Pathway with "Fast-Track"
- Postoperative Usual Protocol (Active Comparator): The postoperative time and the clinical cares in patients with uncomplicated acute appendicitis, are defined by responsability sugery as he thinks he should be according to the literature.
  Interventions: Other: Postoperative Usual Protocol

INTERVENTIONS:
Other: Clinical Pathway with "Fast-Track" — Care described in the critical pathway during postoperative like the moment when the patients can eat, can move or are discharged.
  Arms: Clinical Pathway With "Fast-Track"
Other: Postoperative Usual Protocol — Cares step by step as sugery responsable thinks are the best for patients until discharge.
  Arms: Postoperative Usual Protocol

SUMMARY:
The aim of this study is to reduce the postoperative hospital stay, without increasing morbidity and mortality postoperative, expressed in terms of rate of complications and readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with uncomplicated acute appendicitis urgently.
* Signing the consent of participation and commitment to attend reviews.

Exclusion Criteria:

* Suspected liver disease.
* Coagulation disorders.
* Patients in septic shock.
* Pregnant patients.
* Patients with symptoms compatible with acute uncomplicated appendicitis (plastron appendix, perforated appendicitis or diffuse peritonitis), or had 5 to more days of evolution).
* No sign consent for participation in it.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative Hospital Stay | From the first moment after surgery within 3 months
  Measure the time from when the patient leaves the operating room until discharge

SECONDARY OUTCOMES:
Overall satisfaction (Study the degree of satisfaction that the patient has received assistance as) | From the first moment after surgery within 3 months
  Study the degree of satisfaction that the patient has received assistance as

CONTACTS AND LOCATIONS:
Overall Officials: Juan A. Luján Mompean, Study Director — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Hospital Universitario Virgen de La Arrixaca, Murcia, Murcia, Spain